CLINICAL TRIAL: NCT01184378
Title: Study of Tolerance and Lipid Digestibility of a Formula in Healthy 3 Months Infants
Brief Title: Tolerance and Digestibility of a New Formula in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lactalis (Industry)
Responsible Party: Pascale le Ruyet PhD, Lactalis RetD
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LRD-08-15
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Steatorrhea; Growth
Keywords: infant formula; dairy fat; soluble milk protein
MeSH Terms: conditions — Steatorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control formula (Placebo Comparator): formula containing only vegetable fats
  Interventions: Dietary Supplement: dairy lipids and soluble milk proteins
- new formula (Experimental): new formula with dairy lipids and soluble milk proteins
  Interventions: Dietary Supplement: dairy lipids and soluble milk proteins

INTERVENTIONS:
Dietary Supplement: dairy lipids and soluble milk proteins — one month formula supplementation feces are collected during a 3 days period after 15 and 30 days of formula intake

SUMMARY:
The great majority of infants formula contain fats exclusively from vegetable oil. Nevertheless, the use of both vegetable and dairy lipids is on a real interest to obtain an infant formula closer to the nutritional composition of maternal milk.

ELIGIBILITY:
Inclusion Criteria:

* normal growth;
* considered as healthy by the investigator according to the medical interrogation and the clinical examination;
* receiving exclusively infant formula for at least 15 days.
* without any solid food during the month of the study

Exclusion Criteria:

* Premature born children or small born weights;
* Children breast-fed or weaned for less than 15 days;
* Children with solid food
* Food allergy, particularly in milk proteins allergy , and lactose intolerance ;
* Tumoral, inflammatory, cardiac, lung, renal, digestive diseases(syndrome of malabsorption);
* Digestive pathology previous to the inclusion, in particular infectious (rotavirus, gastroenteritis) or functional symptoms (important stomach pains, colicky) having required a lot of change in formula quality;
* Children under medical treatment (ex: paracetamol).

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
digestibility of lipids in formula | during the 30d consumption period
  lipid content determination in feces during a 3 days period of collection after 15d and 30d of formula intake

SECONDARY OUTCOMES:
tolerance and growth | during the 30d of formula intake

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Faculté de Médecine, Dijon
  - Hopital Mère-Enfants, Rennes